CLINICAL TRIAL: NCT05007717
Title: Data-informed Stepped Care (DiSC) to Improve Adolescent HIV Outcomes (UH3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Pamela Kohler, Associate Professor: School of Nursing; Associate Professor: Public Health/Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: STUDY00011096; UH3HD096906 (NIH)
Record Dates: First submitted 2021-07-13; First posted 2021-08-16 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Adolescent Behavior; Hiv
Keywords: stepped care
MeSH Terms: conditions — Adolescent Behavior; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Data-informed Stepped Care (DiSC) arm (Experimental): At intervention sites, HCW will assign ALHIV to different levels or intensity of HIV services depending on their current and anticipated health care needs. The stepped care framework is designed to be flexible, to accommodate variable individual and social support services available at each facility.
  Interventions: Behavioral: Data-informed Stepped Care (DiSC)
- Standard of care (No Intervention): Sites randomized to the control arm will continue with standard of care approaches for adolescent clinic visits (usually 1-3 monthly visits) regardless of health care needs and additional support as needed.

INTERVENTIONS:
Behavioral: Data-informed Stepped Care (DiSC) — The DiSC intervention is comprised of a data-driven system to assign adolescents to care based on their health needs and the different levels of care for each assignment group.
  The trajectory of services moves from a relative position of ALHIV autonomy to more intensive service provision. Intervention steps start with 1) multi-month refills or community treatment delivery (differentiated care); 2) a standard of care level for those with medical needs such as pregnancy or opportunistic infections or patient choice; 3) patient reminders/tracking and counseling and referral services for mental health needs; 4) case management of unsuppressed individuals, including enhanced counseling and case conference problem-solving
  Arms: Data-informed Stepped Care (DiSC) arm

SUMMARY:
The investigators will conduct a Phase III cluster randomized controlled trial (cRCT) to evaluate the effectiveness of the implementation of a data-informed stepped care (DiSC) intervention for HIV treatment management among adolescents living with HIV (ALHIV) in high-volume HIV clinics in Kenya. The DiSC intervention is comprised of a system to assign ALHIV to care based on their health needs and the different levels of care for each assignment group. The primary outcome will be ALHIV retention, and the secondary outcomes will include adherence, viral non-suppression, and receipt of differentiated care among ALHIV.

DETAILED DESCRIPTION:
UNAIDS '95-95-95' targets cannot be achieved without additional support for adolescents living with HIV (ALHIV) to increase retention in care and to support viral suppression. Risk prediction tools as well as a stepped care approach to care can support differentiation of ALHIV to different risk groups, and tailor care based on risk.

The investigators have conducted informative work with ALHIV, caregivers, healthcare workers (HCW) and policy makers, and has developed a clinical prediction tool to identify ALHIV at highest risk of not being retained in care and poor viral suppression that could be adapted to identify adolescents who may need more support in their care. Understanding how best to use the risk prediction tool as well as how to tailor services based on risk may ultimately result in more efficient HIV care services, as well as adequate support for ALHIV at highest risk of poor outcomes.

Building on that informative work, in this protocol, the investigators will conduct a Phase III cluster randomized controlled trial (cRCT) by implementing a data-informed stepped care (DiSC) intervention of ALHIV HIV treatment management in high-volume HIV clinics in Kenya.

The cRCT will be conducted at up to 24 HIV care and treatment facilities located in Kisumu, Homabay, Migori county in Western Kenya, in which approximately 2000 HIV positive adolescents and young adults ages 10-24 years enrolled in HIV care will be recruited in this study.

Clinics randomized to the DiSC intervention arm will use a data-driven system to assign ALHIV to different levels of care depending on their current and anticipated health care needs. The intervention will be delivered at the individual level by HCW providing routine care during routine HIV clinic visits. Clinics randomized to the control arm will continue with standard of care approaches for adolescent clinic visits (usually 1-3 monthly visits), regardless of health care needs and additional support as needed.

As secondary objectives, this study also aims to evaluate the effectiveness of the DiSC intervention on ALHIV cascade outcomes (adherence, viral non-suppression) and receiving differentiated HIV care based on health status evaluation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Enrolled in HIV care
* Provision of informed consent
* Willing and able to give informed consent

Exclusion Criteria:

- Not able or willing to give informed consent

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1911 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Kohler, RN, MPH, PhD, Principal Investigator — University of Washington
Locations (24):
- Kenya (24):
  - Asumbi Health Centre, Homa Bay
  - Homa Hills Health Centre, Homa Bay
  - Kendu Adventist Hospital, Homa Bay
  - Marindi Sub County Referral Hospital, Homa Bay
  - Mbita District Hospital, Homa Bay
  - Rachuonyo District Hospital, Homa Bay
  - Rangwe Sub-District Hospital, Homa Bay
  - Shirikisho Health Centre, Homa Bay
  - Suba District Hospital, Homa Bay
  - Nyabondo Mission Hospital, Kisumu
  - Nyahera Sub County Hospital, Kisumu
  - Nyang'oma Health Centre, Kisumu
  - Rabour Health Centre, Kisumu
  - St. Elizabeth Chiga, Kisumu
  - Awendo Sub County Hospital, Migori
  - Dede Health Centre, Migori
  - Godkwer, Migori
  - Macalder Mission Hospital, Migori
  - Migori County Mission Hospital, Migori
  - Nyamaraga Health Centre, Migori
  - Rongo Sub County Hospital, Migori
  - Sony Medical Centre, Migori
  - St. Joseph's Mission Hospital, Migori
  - Uriri Sub County Hospital, Migori

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all IPD that underlie results in the primary publication after deidentification procedures.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: The final public-facing repository for clinical data and/or biospecimen information will be the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH)
URL: https://dash.nichd.nih.gov

REFERENCES:
- [Derived] Chhun N, Mangale DI, Agot K, Owade WA, Kadima J, Badia J, Kibugi JK, Kohler PK, John-Stewart G, Beima-Sofie K. Determinants of implementation of a stepped care intervention for adolescents and youth living with HIV in Kenya: a qualitative evaluation. BMC Health Serv Res. 2025 May 15;25(1):702. doi: 10.1186/s12913-025-12875-7. PMID 40369586
- [Derived] Kohler P, Agot K, Njuguna IN, Dyer J, Badia J, Jiang W, Beima-Sofie K, Chhun N, Inwani I, Shah SK, Richardson BA, Chaktoura N, John-Stewart G. Data-informed stepped care to improve youth engagement in HIV care in Kenya: a protocol for a cluster randomised trial of a health service intervention. BMJ Open. 2022 Oct 31;12(10):e062134. doi: 10.1136/bmjopen-2022-062134. PMID 36316073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 24 HIV care and treatment facilities located in Western Kenya between April 2022 and July 2022. The first participant was enrolled on April 19, 2022 and the last participant was enrolled on July 19, 2022.
Pre-assignment Details: The intervention was implemented at clinic-level, then people at clinics were recruited for participation. Participants at the intervention sites received the intervention; participants at the control sites received standard of care.
Units Other Than Participants: facility
Groups:
- Data-informed Stepped Care (DiSC) Arm: Participants at intervention facilities received different levels or intensity of HIV services depending on their current and anticipated health care needs.
  Data-informed Stepped Care (DiSC): The DiSC intervention is comprised of a data-driven system to assign adolescents to care based on their health needs and the different levels of care for each assignment group.
  The trajectory of services moves from a relative position of ALHIV autonomy to more intensive service provision. Intervention steps start with 1) multi-month refills or community treatment delivery (differentiated care); 2) a standard of care level for those with medical needs such as pregnancy or opportunistic infections or patient choice; 3) patient reminders/tracking and counseling and referral services for mental health needs; 4) case management of unsuppressed individuals, including enhanced counseling and case conference problem-solving
- Standard of Care: Participants at the control facilities continued with standard of care approaches for adolescent clinic visits (usually 1-3 monthly visits) regardless of health care needs and additional support as needed.
Period: Overall Study
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care
Started | 895; 12 facility | 1016; 12 facility
Completed | 892; 12 facility | 1014; 12 facility
Not Completed | 3; 0 facility | 2; 0 facility
Not completed — Death | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Data-informed Stepped Care (DiSC) Arm: Participants at intervention sites received different levels or intensity of HIV services depending on their current and anticipated health care needs.
  Data-informed Stepped Care (DiSC): The DiSC intervention is comprised of a data-driven system to assign adolescents to care based on their health needs and the different levels of care for each assignment group.
  The trajectory of services moves from a relative position of ALHIV autonomy to more intensive service provision. Intervention steps start with 1) multi-month refills or community treatment delivery (differentiated care); 2) a standard of care level for those with medical needs such as pregnancy or opportunistic infections or patient choice; 3) patient reminders/tracking and counseling and referral services for mental health needs; 4) case management of unsuppressed individuals, including enhanced counseling and case conference problem-solving
- Standard of Care: Participants at the control sites continued with standard of care approaches for adolescent clinic visits (usually 1-3 monthly visits) regardless of health care needs and additional support as needed.
- Total: Total of all reporting groups
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care | Total
Number analyzed (Participants) | 895 | 1016 | 1911
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Seven participants missed the behavioral survey at baseline.
  years
    number analyzed (Participants) | 888 | 1016 | 1904
    (all) | 16 [14 to 19] | 17 [15 to 19] | 17 [14 to 19]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Seven participants missed the behavioral survey at baseline. Six participants reported unknown or no answer
  Participants
    number analyzed (Participants) | 885 | 1013 | 1898
    Female | 532 | 570 | 1102
    Male | 353 | 443 | 796
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 895 | 1016 | 1911
Always come to this clinic by yourself [Count of Participants; unit: Participants] — Population: Seven participants missed the behavioral survey at baseline. Seven participants reported unknown or no answer.
  Participants
    number analyzed (Participants) | 886 | 1011 | 1897
    (all) | 541 | 694 | 1235

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Missed Visits
Description: We will evaluate retention using a definition of missed visit and calculate the proportion of scheduled visits that are missed. Missed visits will be defined as a participant not seen within 30 days after each scheduled visit. Each scheduled visit will be classified as missed versus not missed.
Time Frame: 12 months
Population: Five participants did not have clinic visit data matched in the medical records.
Measure: Count of Units; unit: Scheduled visits
Units Other Than Participants: Scheduled visits
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care
Number analyzed (Participants) | 892 | 1014
Number analyzed (Scheduled visits) | 4784 | 5248
Scheduled visits | 406 | 433
Statistical Analysis 1: Comparison: Data-informed Stepped Care (DiSC) Arm vs Standard of Care; Test type: Superiority; p = 0.631, Mixed Models Analysis; Adjusted for ever missing a visit during a 6 months pre-enrollment period and always coming to clinic by yourself; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.89 to 1.20]

2. Secondary Outcome: Proportion of Viral Load Results Showing Viral Non-suppression
Description: We will evaluate viral load test results and calculate the proportion of results that show non-suppression. Viral non-suppression will be defined as having HIV RNA viral loads (VL) >1,000 copies per milliliter. Each VL test result will be classified as VL suppressed vs. unsuppressed.
Time Frame: 12 months
Population: One hundred and forty-four participants did not have viral loads data matched in the medical records.
Measure: Count of Units; unit: Viral load assays
Units Other Than Participants: Viral load assays
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care
Number analyzed (Participants) | 833 | 934
Number analyzed (Viral load assays) | 1624 | 1899
Viral load assays | 125 | 184
Statistical Analysis 1: Comparison: Data-informed Stepped Care (DiSC) Arm vs Standard of Care; Test type: Superiority; p = 0.237, Mixed Models Analysis; Adjusted for ever being virally unsuppressed during a 6 months pre-enrollment period and always coming to clinic by yourself; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.54 to 1.16]

3. Secondary Outcome: Proportion of Visit Intervals With Good Adherence
Description: We will evaluate adherence by calculating the number of pills dispensed divided by the number of days during an inter-visit interval. A proportion of adherence greater than 0.8 will be classified as good adherence. The level of adherence during the past inter-visit interval will be assessed at each visit.
Time Frame: 12 months
Population: Seven participants did not have clinic visit data matched in the medical records.
Measure: Count of Units; unit: Intervals
Units Other Than Participants: Intervals
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care
Number analyzed (Participants) | 891 | 1013
Number analyzed (Intervals) | 4382 | 4741
Intervals | 4065 | 4486
Statistical Analysis 1: Comparison: Data-informed Stepped Care (DiSC) Arm vs Standard of Care; Test type: Superiority; p = 0.386, Mixed Models Analysis; Adjusted for always having >80% coverage during a 6 months pre-enrollment period and always coming to clinic by yourself; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.94 to 1.02]

4. Secondary Outcome: Incidence Rate of Loss to Follow-up
Description: We will also analyze retention using loss to follow-up (LTFU). LTFU will be defined as a participant not seen within 30 days of a scheduled visit and not return to care within the 12-month study period. The incidence rate of LTFU is the ratio of the number of new cases of LTFU to the total time the study participants was at risk of LTFU. The denominator is the sum of the time each participant (person-year) was observed, totaled for all participants.
Time Frame: 12 months
Population: Five participants did not have clinic visit data matched in the medical records.
Measure: Count of Units; unit: Person-year
Units Other Than Participants: Person-year
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care
Number analyzed (Participants) | 892 | 1014
Number analyzed (Person-year) | 796 | 913
Person-year | 61 | 73
Statistical Analysis 1: Comparison: Data-informed Stepped Care (DiSC) Arm vs Standard of Care; Test type: Superiority; p = 0.991, Regression, Cox; Adjusted for always coming to clinic by yourself; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.71 to 1.41]

5. Secondary Outcome: Proportion of Visits Enrolled in Differentiated Care Services (Fast-track Visits)
Description: We will calculate the proportion of visits enrolled in differentiated care using two definitions. The first is fast-track visit, which evaluates if participants are assigned to fast-track status during visits. Each visit will be assessed as enrolled in differentiated care (assigned to fast-track) or not.
Time Frame: 12 months
Population: Five participants did not have clinic visit data matched in the medical records.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care
Number analyzed (Participants) | 892 | 1014
Number analyzed (Visits) | 4586 | 4963
Visits | 517 | 520
Statistical Analysis 1: Comparison: Data-informed Stepped Care (DiSC) Arm vs Standard of Care; Test type: Superiority; p = 0.037, Mixed Models Analysis; Adjusted for having been given fast track visits during a 6 months pre-enrollment period and always coming to clinic by yourself; Risk Ratio (RR) = 1.21, 95% CI 2-sided [1.01 to 1.46]

6. Secondary Outcome: Proportion of Visits Enrolled in Differentiated Care Services (Multi-month Refills)
Description: We will calculate the proportion of visits enrolled in differentiated care using two definitions. The second is multi-month prescription refills, which evaluates if participants are given multi-month refill intervals more than 3 months. Each visit will be assessed as enrolled in differentiated care (given multi-month refills) or not.
Time Frame: 12 months
Population: Five participants did not have clinic visit data matched in the medical records.
Measure: Count of Units; unit: Scheduled visits
Units Other Than Participants: Scheduled visits
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care
Number analyzed (Participants) | 892 | 1014
Number analyzed (Scheduled visits) | 5273 | 5760
Scheduled visits | 1939 | 2180
Statistical Analysis 1: Comparison: Data-informed Stepped Care (DiSC) Arm vs Standard of Care; Test type: Superiority; p = 0.276, Mixed Models Analysis; Adjusted for having been given long intervals during a 6 months pre-enrollment period and always coming to clinic by yourself; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.97 to 1.12]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Data-informed Stepped Care (DiSC) Arm | Standard of Care
All-Cause Mortality (participants affected / at risk) | 3/895 | 2/1016
Serious Adverse Events (participants affected / at risk) | 1/895 | 0/1016
Other Adverse Events (participants affected / at risk) | 0/895 | 0/1016
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Data-informed Stepped Care (DiSC) Arm (N=895) | Standard of Care (N=1016)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | NA — Complained of ringing in the ears, worsened and eventually lost hearing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT05007717/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT05007717/SAP_001.pdf